CLINICAL TRIAL: NCT03687905
Title: Comparative Study Between Chloroquine and Hydroxychloroquine as Therapeutic Modalities for Children and Adolescents With Proliferative Lupus Nephritis
Brief Title: Proliferative Lupus Nephritis Treatment With Chloroquine and Hydroxychloroquine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Fatma Sayed Ahmed Gheet, Resident Pediatercian, Tanta University
Other Study IDs: Fatma
Record Dates: First submitted 2018-09-18; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Proliferative Nephritis; Chloroquine Retinopathy
MeSH Terms: interventions — Chloroquine; Hydroxychloroquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lupus nephritis III or IV/chloroquine: receiving chloroquine with daily dose 5 mg/kg
  Interventions: Drug: Chloroquine
- Lupus nephritis III or IV/hydroxychloroquine: receiving hydroxycholorquine with daily dose 5 mg/kg
  Interventions: Drug: Hydroxychloroquine
- Systemic lupus erythematosus: not received hydroxychloroquine nor chloroquine .

INTERVENTIONS:
Drug: Chloroquine — group1 received chloroquine .
  Other Names: alexoquine
  Groups: Lupus nephritis III or IV/chloroquine
Drug: Hydroxychloroquine — Group 2 received hydroxychloroquine
  Other Names: hydroquine
  Groups: Lupus nephritis III or IV/hydroxychloroquine

SUMMARY:
Evaluation the efficacy of chloroquine and hydroxychloroquine in the treatment of proliferative lupus nephritis class III and IV in children and adolescents and evaluate the side effects of both drugs .

DETAILED DESCRIPTION:
All patients will fulfill the diagnostic criteria of SLE. The diagnosis of systemic lupus erythematosus is based on clinical and laboratory criteria. The criteria set developed by the American College of Rheumatology (ACR) and diagnosed wih lupus nephritis class III and IV .

Inclusion Criteria:

* Children and adolescents who fulfill diagnostics criteria of SLE and diagnosed with lupus nephritis class III and IV.
* All patients will be received steroids , MMF and Angiotensin Converting Enzyme.

Exclusion Criteria:

* Patients diagnosed with lupus nephritis class I,II,V and VI.
* Patients received Cyclophosphamide in stead of MMF.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents who fulfill diagnostics criteria of SLE and diagnosed with lupus nephritis class III and IV.
* All patients will be received steroids , MMF and Angiotensin Converting Enzyme.

Exclusion Criteria:

* Patients diagnosed with lupus nephritis class I,II,V and VI.
* Patients received Cyclophosphamide in stead of MMF.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: • All patients will fulfill the diagnostic criteria of SLE. The diagnosis of systemic lupus erythematosus is based on clinical and laboratory criteria. The criteria set developed by the American College of Rheumatology (ACR) and diagnosed wih lupus nephritis class III and IV
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Fundus examination as screening test | 12 months
  Detection of chloroquine and hydroxychloroquine related retinal toxicity at early stage.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma S Gheet, M.B.,BCh, Principal Investigator — Tanta University
Locations (1):
- Fatma Gheet, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data is secret.

REFERENCES:
- [Derived] Gheet FS, Dawoud HE, El-Shahaby WA, Elrifaey SM, Abdelnabi HH. Hydroxychloroquine in children with proliferative lupus nephritis: a randomized clinical trial. Eur J Pediatr. 2023 Apr;182(4):1685-1695. doi: 10.1007/s00431-023-04837-0. Epub 2023 Feb 8. PMID 36752895